CLINICAL TRIAL: NCT02540772
Title: Study of the Neuroanatomical Circuits, Predictors and Prognostic Factors of Spontaneous Confabulation: Designing an Assessment and Rehabilitation Program
Brief Title: Neuropsychological Rehabilitation of Spontaneous Confabulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Triviño Mosquera (Other)
Responsible Party: Sponsor-Investigator, Monica Triviño Mosquera, Psychology PhD, San Rafael University Hospital, Granada, Spain
Organization: San Rafael University Hospital, Granada, Spain (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Conf-01
Record Dates: First submitted 2015-08-15; First posted 2015-09-04 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Memory Disorders
Keywords: Confabulations; Neuropsychological rehabilitation; Memory
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuropsychological treatment (Experimental): The tested treatment is a combination of neuropsychological rehabilitation procedures: learning, episodic memory recall after a delay, selective attention, inhibition of predominant responses and awareness of deficits.
  Interventions: Behavioral: Neuropsychological treatment
- No treatment (No Intervention): Patients in the control group only performed the baselines.

INTERVENTIONS:
Behavioral: Neuropsychological treatment — Participants had to learn some brief material (words, faces, pictures, news), after which they were asked for an immediate and a delayed recall. After both recalls, participants were confronted with feedback about correct responses, non-responses and errors (i.e., confabulations and errors of attribution). This type of feedback worked on: 1) selective attention during the learning phase, training patients to focus on the relevant details of the stimuli; 2) monitoring processes during the retrieval phase, reinforcing the strategic search and training patients to inhibit traces that were irrelevant; and 3) memory control processes after the retrieval phase. The treatment consisted of 9 sessions and lasted for 3 weeks and the participants performed a baseline before and after treatment.
  Other Names: Confabulations treatment
  Arms: Neuropsychological treatment

SUMMARY:
Confabulators consistently generate false memories without intention to deceive and with great feeling of rightness. However, there is currently no known effective treatment for them. In order to fill this gap, the aim of this trial was to design a neuropsychological treatment based on the current theoretical models and test it experimentally in two groups of confabulators: experimental vs. control. The treatment consisted of some brief material that patients had to learn and recall at both immediate and delayed moments. After both recollections, patients were given feedback about their performance (errors and correct responses). Pre-treatment and post-treatment baselines were administered. Confabulators in the control group performed the baselines without treatment, and were then offered the treatment after the second baseline.

ELIGIBILITY:
Inclusion Criteria:

* The presence of spontaneous confabulations after acute brain injury, for at least three months and without clinical improvement (interfering with the patient's daily life with frequent arguments and exhaustive supervision).
* The presence of momentary confabulations in the Spanish adaptation of Dalla Barba provoked confabulation interview.
* Prior to injury, all patients should be completely independent for daily living.

Exclusion Criteria:

* The presence of impairment in alertness.
* Dementia.
* Acute confusional state.
* A history of alcohol or drug abuse.
* Psychiatric antecedents.

Ages: 35 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Triviño, PhD, Principal Investigator — San Rafael University Hospital
Locations (1):
- San Rafael University Hospital, Granada, Granada, Spain

REFERENCES:
- [Background] Gilboa A, Alain C, Stuss DT, Melo B, Miller S, Moscovitch M. Mechanisms of spontaneous confabulations: a strategic retrieval account. Brain. 2006 Jun;129(Pt 6):1399-414. doi: 10.1093/brain/awl093. Epub 2006 Apr 25. PMID 16638795
- [Background] Moscovitch M, Melo B. Strategic retrieval and the frontal lobes: evidence from confabulation and amnesia. Neuropsychologia. 1997 Jul;35(7):1017-34. doi: 10.1016/s0028-3932(97)00028-6. PMID 9226662
- [Background] Schnider A. The confabulating mind. How the brain creates reality. Oxford: Oxford University Press; 2008.
- [Background] Nahum L, Bouzerda-Wahlen A, Guggisberg A, Ptak R, Schnider A. Forms of confabulation: dissociations and associations. Neuropsychologia. 2012 Aug;50(10):2524-34. doi: 10.1016/j.neuropsychologia.2012.06.026. Epub 2012 Jul 7. PMID 22781813
- [Background] Ciaramelli E, Ghetti S, Borsotti M. Divided attention during retrieval suppresses false recognition in confabulation. Cortex. 2009 Feb;45(2):141-53. doi: 10.1016/j.cortex.2007.10.006. Epub 2008 Feb 6. PMID 19150516
- [Background] Dayus B, Van den Broek MD. Treatment of stable delusional confabulations using self-monitoring training. Neuropsychol Rehabil, 2000; 10(4):415-427.
- [Background] Del Grosso Destreri N, Farina E, Calabrese E, Pinardi G, Imbornone E, Mariani C. Frontal impairment and confabulation after herpes simplex encephalitis: A case report. Arch Phys Med Rehabil. 2002 Mar;83(3):423-6. doi: 10.1053/apmr.2002.29646. PMID 11887126
- [Background] Dalla Barba G, Decaix C. "Do you remember what you did on March 13, 1985?" A case study of confabulatory hypermnesia. Cortex. 2009 May;45(5):566-74. doi: 10.1016/j.cortex.2008.03.009. Epub 2008 Jun 5. PMID 18621364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited during the period between April 2013 and April 2015 at the San Rafael Hospital where they were admitted for rehabilitation after acquired brain injury.
Pre-assignment Details: Due to the absence of confabulations in the Dalla Barba interview two participants were excluded. Another two participants were excluded because a deficit in alertness.
Groups:
- Neuropsychological Treatment: The tested treatment is a combination of neuropsychological rehabilitation procedures: learning, episodic memory recall after a delay, selective attention, inhibition of predominant responses and awareness of deficits.
  Neuropsychological treatment: Participants had to learn some brief material (words, faces, pictures, news), after which they were asked for an immediate and a delayed recall. After both recalls, participants were confronted with feedback about correct responses, non-responses and errors. This type of feedback worked on: 1) selective attention during the learning phase, training patients to focus on the relevant details of the stimuli; 2) monitoring processes during the retrieval phase, reinforcing the strategic search and training patients to inhibit traces that were irrelevant; and 3) memory control processes after the retrieval phase. The treatment consisted of 9 sessions and lasted for 3 weeks and the participants performed a baseline before and after treatment.
Period: Overall Study
Arm/Group | Neuropsychological Treatment | No Treatment
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Minimum number for comparison of means
Groups:
- Neuropsychological Treatment: Combination of neuropsychological rehabilitation procedures: learning, episodic memory recall after a delay, selective attention, inhibition of predominant responses and awareness of deficits.
- Total: Total of all reporting groups
Arm/Group | Neuropsychological Treatment | No Treatment | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (14.3) | 68.1 (11.2) | 66.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Confabulations
Description: The confabulations recorded were 1) guessed answers, 2) confusions in time and space, 3) a mixture of two or more stimuli presented, and 4) devised or bizarre responses.
  Scores ranged from 0 (no confabulations) to unlimited number of them (because devised or bizarre responses were recorded) and consisted of the sum of all the confabulations produced during the baseline. The values in the table represent the mean of confabulations for each group (Neuropsychological treatment or No treatment) in the 3 sessions at each baseline (pre- and post-treatment).
Time Frame: Measures were recorded during 3 sessions administered in 1 week before (pre-baseline) and during 3 sessions after the treatment (post-baseline). In the control group, pre and post baselines were also recorded but without any treatment between them
Population: We used preliminary data from the first 5 patients using the G*Power software to calculate the sample size. From them, to detect differences through a Student t-test considering the significance level is 5%, the sample size was estimated in 7 subjects per group with an alpha of 0.95. We expanded to 10 to ensure greater power.
Measure: Mean (Standard Deviation); unit: Confabulations
Arm/Group | Neuropsychological Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
Confabulations
  Pre baseline | 30.0 (9.9) | 29.9 (13.8)
  Post baseline | 8.1 (4.2) | 35.5 (11.3)

2. Primary Outcome: Number of Correct Responses
Description: Scores ranged from 0 (no correct answers) to 72 (12 stimuli remembered twice in each session: firstly, in a immediate recall after learning, and secondly, in a delayed recall after 10 minutes).
  The values in the table represent the mean of correct responses for each group (Neuropsychological treatment or No treatment) in the 3 sessions at each baseline (pre- and post-treatment).
Time Frame: as for outcome 1
Population: Minimum number for comparison of means calculated with G*Power software (see Analysis Population Description of previous outcome measure data, i.e., confabulations).
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Neuropsychological Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
Correct responses
  Pre baseline | 22.0 (13.6) | 20.9 (10.6)
  Post baseline | 42.6 (18.7) | 22.0 (8.9)

3. Primary Outcome: Number of Non-responses
Description: Scores ranged from 0 (no non-responses) to 72 (12 stimuli remembered twice in each session: firstly, in a immediate recall after learning, and secondly, in a delayed recall after 10 minutes).
  The values in the table represent the mean of non-responses for each group (Neuropsychological treatment or No treatment) in the 3 sessions at each baseline (pre- and post-treatment).
Time Frame: as for outcome 1
Population: Minimum number for comparison of means calculated with G*Power software (see Analysis Population Description of the first outcome measure data, i.e., confabulations).
Measure: Mean (Standard Deviation); unit: Non-responses
Arm/Group | Neuropsychological Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
Non-responses
  Pre baseline | 26.3 (15.8) | 29.5 (11.8)
  Post baseline | 22.3 (17.5) | 19.2 (8.8)

4. Secondary Outcome: Number of Errors in Source Attribution
Description: After the recall of the material, patients were also asked to remember which modality corresponded to each recall (i.e., seen, heard or imagined), and who had presented the material during the learning session (i.e., the therapist or themselves).
  Scores ranged from 0 (if all answers were non-responses) to unlimited number (depending on number of confabulations produced by patients).
  The values in the table represent the mean of errors in source attribution for each group (Neuropsychological treatment or No treatment) in the 3 sessions at each baseline (pre- and post-treatment).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Errors in source attribution
Arm/Group | Neuropsychological Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
Errors in source attribution
  Pre baseline | 25.1 (6.1) | 25.7 (12.5)
  Post baseline | 12.2 (7.0) | 30.2 (11.6)

ADVERSE EVENTS:
Time Frame: One week
Description: A neuropsychological assessment and an interview to the relatives were administered before and after treatment to ensure that the treatment did not produce undesired effects on cognition (worsening of the confabulations) or behavior (severe behavioral disorders) in the patients. This assessment was administered in 3 sessions over a week.
Arm/Group | Neuropsychological Treatment | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 7/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuropsychological Treatment (N=10) | No Treatment (N=10)
Worsening of confabulations (Nervous system disorders) | 0 (0) | 7 (7) — Number of confabulations in the Dalla Barba provoked confabulation interview
Worsening of Behavioral Disorders (Nervous system disorders) | 0 (0) | 0 (0) — Increased confusional state and escapism. Interview to relatives.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuropsychological Treatment (N=10) | No Treatment (N=10)
Worsening of memory (Nervous system disorders) | 0 (0) | 0 (0) — Memory execution in a memory test (Test Aprendizaje Verbal España Complutense, as a version of the California Verbal Learning test)
Worsening of attention (Nervous system disorders) | 0 (0) | 0 (0) — Worsening in selective attention in neuropsychological test: Picture Completion (WAIS-III)
Worsening of working memory (Nervous system disorders) | 0 (0) | 0 (0) — Worsening of working memory in neuropsychological tests: digit span (WAIS-III) and spatial span (WMS-III)
Worsening of executive functions (Nervous system disorders) | 0 (0) | 0 (0) — Worsening of fluency, planning and reasoning in different neuropsychological tests: animal fluency, Key Search (BADS), Similarities (WAIS-III)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No